CLINICAL TRIAL: NCT02688023
Title: A Pilot Phase II Study of Triplet Chemotherapy Regimen in Neoadjuvant Chemotherapy of Patients With Resectable Colorectal Cancer
Brief Title: Neoadjuvant Triplet Chemotherapy Regimen in Patients With Resectable Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Huang, MD PhD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-052
Record Dates: First submitted 2016-02-11; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Cancer
Keywords: 5-fluorouracil; Irinotecan; Oxaliplatin; Colorectal cancer; neoadjuvant; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm Irinotecan-Oxaliplatin-5-Fluorouracil/leucovorin (Experimental): Irinotecan,oxaliplatin and 5-fluorouracil/leucovorin(5-fluorouracil/leucovorin can be substituted with Capecitabine or S-1)
  Interventions: Drug: oxaliplatin;irinotecan;leucovorin;5-fluorouracil;capecitabine;S-1

INTERVENTIONS:
Drug: oxaliplatin;irinotecan;leucovorin;5-fluorouracil;capecitabine;S-1 — The regimen consisted of irinotecan 150mg/m2 administered as an intravenous infusion on day 1, oxaliplatin 85 mg/m2 administered intravenously on day 2, leucovorin 200 mg intravenously on day 2, 5-fluorouracil 500 mg administered by intravenous bolus,followed by 2400 mg/m2 by 44 h continuous intravenous infusion starting on day 2. S-1 (40-60mg orally twice per day for 10 days) or capecitabine (1000mg/m2 orally twice per day for 10 days) can be substituted for intravenous 5-fluorouracil.14 days as a cycle, up to 4 cycles.

SUMMARY:
Colorectal cancer is an aggressive malignancy with a poor overall outcome. The purpose of this study is to evaluate the feasibility, safety and efficacy of neoadjuvant oxaliplatin, irinotecan combined with 5-fluorouraci/leucovorin or S-1 or capecitabine in patients with resectable colorectal cancer.

DETAILED DESCRIPTION:
This is a single arm, phase 2 study of neoadjuvant triplet chemotherapy regimen of oxaliplatin, irinotecan combined with 5-fluorouraci/leucovorin or S-1 or capecitabine in patients with resectable colorectal cancer.Fifty patients will be enrolled in this trial. The primary objective of this study is to determine the 3-year disease-free survival of the patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified colorectal cancer
* clinical stage T4N0-2M0、cT1-3N2M0 or M1(liver metastases only)
* age: 18-70 years
* ECOG 0-2
* adequate bone marrow, liver, renal and cardiac function (no history of ischemic heart disease)
* no prior cancer and/or chemotherapy
* signed informed consent

Exclusion Criteria:

* patients with a history of prior malignancy
* pregnant or lactating patients
* known or suspected brain metastasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 5 years

SECONDARY OUTCOMES:
objective response rate | 2 years
Surgical complete resection rate (R0) | 2 years
overall survival | 6 years
Number of participants with adverse events that are related to treatment | 2 years
Number of participants with surgery complications | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, M.D., Principal Investigator — Cancer Hospital, CAMS
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China